CLINICAL TRIAL: NCT05866341
Title: Influence of the Regular Consumption of a Nitrate Containing Juice Beverage on Gingival Inflammation and the Salivary Nitrate/Nitrite Relationship in Periodontitis Patients
Brief Title: Nitrate Consumption and Gingival Inflammation
Acronym: NITGIN14
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yvonne Jockel-Schneider, Prof. Dr. med. dent., Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NITGIN14
Record Dates: First submitted 2023-04-26; First posted 2023-05-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: double blind randomized prospective placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients were allocated using a computer-generated randomization list in blocks of six either to the test or the placebo group. Assignment to a participant number was done according to the chronological order of enrolment in the study. All therapeutic and diagnostic interventions were performed at the Department of Periodontology of the University Hospital of Wuerzburg. All examinations were performed by two experienced, inter- and intra-calibrated periodontists not being involved in patient assignment and hand out of the experimental juices respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich Diet (Active Comparator): Daily consumption of 200 mg nitrate via the consumption of 300 mL of a nitrate-rich lettuce juice beverage.
  Interventions: Dietary Supplement: nitrate-rich lettuce juice
- Nitrate-depleted Diet (Placebo Comparator): Daily consumption of 300 mL of a nitrate-depleted lettuce juice beverage.
  Interventions: Dietary Supplement: nitrate-depleted lettuce juice

INTERVENTIONS:
Dietary Supplement: nitrate-rich lettuce juice — Consumption of a daily dosage of 200 mg nitrate via the consumption of a 300mö of a nitrate-rich lettuce juice
  Arms: Nitrate-rich Diet
Dietary Supplement: nitrate-depleted lettuce juice — Daily consumption of 300 ml of a nitrate-depleted lettuce juice
  Arms: Nitrate-depleted Diet

SUMMARY:
The aim of this investigation is to evaluate the impact of the 14- day consumption of a nitrate-rich diet on the the extent of gingival inflammation in a cohort of periodontal aftercare patients. Recorded parameters were gingival index, plaque control record, salivary nitrate/nitrite level and vascular parameters

DETAILED DESCRIPTION:
This investigation evaluated the impact of a nitrate-rich diet on the extent of gingival inflammation in a cohort of periodontal aftercare patients. Forty-four (23 test/21 placebo) periodontal aftercare patients with chronic gingivitis were enrolled. At baseline, gingival index (GI), plaque con- trol record (PCR) and salivary nitrate level (SNL) were recorded, followed by sub- and supragingival debridement. Subsequently, participants were randomly provided with 100 ml bottles of a lettuce juice beverage to be consumed 39 daily over 14 days, containing either a standardized amount of nitrate resulting in an intake of approximately 200 mg nitrate per day (test) or being devoid of nitrate (placebo).

ELIGIBILITY:
Inclusion Criteria:

* number of teeth ≥ 10
* body mass index (BMI) ≥ 24 ≤ 30
* presence of mild to moderate gingivitis (Gingiva Index > category GI 0 ≤ category GI 2) at a minimum of 3 teeth
* history of periodontal disease and inclusion in a regular scheme of supportive periodontal therapy (regularly repeated subgingival biofilm removal 2-4 x/year)

Exclusion Criteria:

* manifestation of severe gingivitis (Gingiva Index = 3) at any tooth
* manifestation of inflammatory oral mucosal diseases other than gingivitis
* xerostomia (salivary flow ≤ 0.1 ml/minute)
* inability for regular oral home care
* known allergies and intolerances to any of the ingredients of the experimental juice beverages
* inability to follow the study protocol due to intellectual or physical handicaps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Gingival Index | Baseline
  Gingival Index will be recorded visually according to the modification of the original GI by Lobene et al.
Gingival Index | Day 14
  Gingival Index will be recorded visually according to the modification of the original

SECONDARY OUTCOMES:
Composition the oral microbiota | Baseline
  The microbial composition of pooled paper point plaque samples taken from the 4 deepest periodontal pockets are assessed by 16 S Genome Sequencing on a genus level
Composition the oral microbiota | Day 14
  The microbial composition of pooled paper point plaque samples taken from the 4 deepest periodontal pockets are assessed by 16 S Genome Sequencing on a genus level
Salivary nitrite level | Baseline
  salivary nitrite level (SNIL) was determined in duplicate by high-performance anion-exchange chromatography with suppressed conductivity detection (HPAEC-CD)
Salivary nitrite level | Day 14
  salivary nitrite level (SNIL) was determined in duplicate by high-performance anion-exchange chromatography with suppressed conductivity detection (HPAEC-CD)
Salivary nitrate level | Baseline
  salivary nitrate level was determined in duplicate by high-performance anion-exchange chromatography with suppressed conductivity detection (HPAEC-CD)
Salivary nitrate level | Day 14
  salivary nitrate level was determined in duplicate by high-performance anion-exchange chromatography with suppressed conductivity detection (HPAEC-CD)
Central blood pressure (systolic pressure, diastolic pressure) | Baseline
  Analysis of central blood pressure by pulse wave analysis using the Arteriograph recording system (TensioMed Ltd, Hungary, software 1.9.9.12).
Central blood pressure (systolic pressure, diastolic pressure) | Day 14
  Analysis of central blood pressure by pulse wave analysis using the Arteriograph recording system (TensioMed Ltd, Hungary, software 1.9.9.12).
Peripheral blood pressure (systolic pressure, diastolic pressure) | Baseline
  Analysis of peripheral blood pressure by pulse wave analysis using the Arteriograph recording system (TensioMed Ltd, Hungary, software 1.9.9.12).
Peripheral blood pressure (systolic pressure, diastolic pressure) | Day 14
  Analysis of peripheral blood pressure by pulse wave analysis using the Arteriograph recording system (TensioMed Ltd, Hungary, software 1.9.9.12).

IPD SHARING:
Plan to Share IPD: Undecided